CLINICAL TRIAL: NCT03253952
Title: PROSPECT ADDITION SCI - A PROSPECTive Study of Autonomic Dynamic Dysfunction to Predict infecTIONs After Spinal Cord Injury
Brief Title: A Study of Autonomic Dynamic Dysfunction to Predict Infections After Spinal Cord Injury.
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jan Schwab, Director of Spinal Cord Medicine, Ohio State University
Other Study IDs: 2016H0369
Record Dates: First submitted 2017-08-09; First posted 2017-08-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Trauma, Spinal Cord; SPINAL Fracture
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traumatic Spinal Cord Injury: Observational study - monitoring immune response and heart rate variability
- Traumatic Spine Fracture, Control Group: Observational study - monitoring immune response and heart rate variability acting as a control group.

SUMMARY:
The study is designed to investigate whether autonomic shifts (dysautonomia, sympatho-vagal instability) that develop after SCI have value in predicting SCI-associated infections (SCI-AI). SCI-AI impair outcomes by (1) reducing the intrinsic neurological recovery potential and (2) increasing mortality. Heart Rate Variability (HRV) data will be tracked in both the time and frequency domains to discriminate between the relative contribution of sympathetic and parasympathetic innervation to changes in HRV. The ability to predict infections will enable novel treatments thereby reducing infection-associated mortality and improving neurological and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute isolated spinal cord injury (AIS A-D) planned for surgical stabilization and decompression, lesion may include more than 1 segment
2. Patients with acute isolated spinal fracture, lesion may include more than 1 segment
3. Legal age of the patient
4. Documented informed consent of the patient

Exclusion Criteria:

1. Non-traumatic spinal cord injury
2. Concomitant traumatic brain injury (TBI) (definition: i) patient with severe TBI (Glasgow Coma Scale ≤ 8) and ii) patients with intracranial pressure monitoring sensors)
3. Neoplasia and/or antineoplastic therapy
4. Pregnancy, lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SCI patients (n=50 subjects), Isolated Spinal fracture patients (n=10)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-29 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sympatho-vagal instability as an identifier for patients at risk for Spinal Cord Injury Associated Infections | At all study time-points for a period of 24hours.
  Determining whether discrete signs of loss of autonomic control (dysautonomia), not meeting defined criteria of full-autonomic dysreflexia, also renders patients "at risk" for developing infections.

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Schwab, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States